CLINICAL TRIAL: NCT05928572
Title: Effect of CGM Initiation Approach on Time in Range in People with Type 2 Diabetes
Brief Title: My Diabetes Study - CGM Initiation Approach & Time in Range
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holly Willis (Other)
Responsible Party: Sponsor-Investigator, Holly Willis, Principal Investigator, HealthPartners Institute
Organization: HealthPartners Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A21-292
Record Dates: First submitted 2023-06-14; First posted 2023-07-03 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes
Keywords: continuous glucose monitor; CGM; nutrition; diet; lifestyle; behavior change
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Nutrition-Focused Approach (NFA) (Experimental): NFA arm participants will receive introduction to CGM from a diabetes care provider with emphasis placed on using the CGM data to adjust food choices. The NFA will encourage food choices that align with evidence-based nutrition recommendations for People with Diabetes (PWD), and that achieve internationally recognized glucose targets (e.g. glucose 70-180 mg/dL, and Time In Range > 70%).
  Interventions: Other: CGM initiation approach
- Self-Directed Approach (SDA) (Active Comparator): The SDA arm participants will receive introduction to the CGM from a diabetes care provider using the CGM manufacturer-provided manuals and resources. The SDA will encourage participants to use the CGM device and apps in the way that feels most useful to them. The SDA is intended to reflect current CGM initiation practices, which focus on technical use of the CGM and a general review of CGM data.
  Interventions: Other: CGM initiation approach

INTERVENTIONS:
Other: CGM initiation approach — Use of a nutrition-focused approach versus a self-directed approach during CGM initiation

SUMMARY:
This study includes two phases. The purpose of Phase 1 of this study is to understand if there is a difference between two ways of introducing a continuous glucose monitor (CGM) to people with type 2 diabetes (T2D). The study will evaluate the effect of using a nutrition-focused approach (NFA) versus a self-directed approach (SDA) during CGM initiation on time in range (TIR) glucose. TIR is the percent of time that someone's glucose is between 70 and 180 mg/dL. It is possible that the approach used to introduce the CGM could impact TIR and other outcomes.

The purpose of Phase 2 of the study is to evaluate the impact of discontinuing CGM for 4 months after the completion of the Phase 1 study intervention on CGM-derived metrics, dietary intake assessment, and patient reported outcomes.

DETAILED DESCRIPTION:
Study Design: This is a non-pivotal, randomized, parallel group, two-arm, prospective study. In Phase 1, this 60-day pilot study will evaluate the effect of a Nutrition-Focused Approach (NFA) versus a Self-Directed Approach (SDA) during CGM initiation in people with T2D. It is hypothesized that the NFA arm will see greater improvement in TIR than the SDA arm, due to the potential for dietary improvements that come from the NFA. To test this hypothesis, participants will be randomized 1:1 to either the NFA or the SDA arm. Participants in each arm complete baseline assessments, an in-person CGM initiation appointment, a remote follow-up appointment, and in-person post-intervention assessments. Difference in changes between baseline and post-intervention periods will be assessed.

Arms: In brief, the NFA arm participants will receive introduction to CGM with emphasis placed on using the CGM data to adjust food choices. The NFA will encourage food choices that align with evidence-based nutrition recommendations for people with diabetes (PWD), and that achieve internationally recognized glucose targets (e.g. glucose 70-180 mg/dL, and TIR > 70%). The SDA arm participants will receive introduction to CGM using manufacturer-provided manuals and resources. The SDA will encourage participants to use the device and apps in the way they feel is most useful to them. The SDA is intended to reflect current CGM initiation practices, which focus on technical use of the CGM and a general review of CGM data.

Intervention: Prior to the intervention, there is an approximately 10-day baseline assessment period, which includes blinded baseline CGM data assessment. The intervention begins on Day 0, which is the day the CGM sensor is paired with apps on the participant's personal cell phone. The intervention follows participants for approximately 50 days, which includes up to 10-days of post-intervention CGM data assessment (approximately Days 40 to 50). During the final 10 days, the participant is instructed to continue using the CGM device in accordance with the guidance provided based on randomization arm.

Sample Size: This study expects to enroll at least N=132 participants with the expectation for an analytic sample size of N=120. This sample size is based on the N needed to adequately power the primary hypothesis with a realistic and clinically meaningful effect size for % TIR.

Phase 2 will evaluate the impact of discontinuing CGM for 4 months after the completion of the Phase 1 study intervention for combined NFA and SDA arms. There is no intervention provided during Phase 2. The sample size is dependent the number of participants that complete Phase 1 and continue through the Phase 2 follow-up assessment period.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years of age
* T2D diagnosis
* HbA1c 7.0%-10.0% based on point-of-care test at screening
* Taking no diabetes medication or taking stable-dose diabetes medication(s) for at least 30 days; willing to maintain stable diabetes medication regimen for the duration of the study
* Has a personal cellular-plan or wifi-connected smartphone that is compatible with required CGM apps and which will be consistently available for duration of the study
* Has not used a personal CGM system within 90 days
* Willing and able to wear CGM and use the associated CGM mobile apps throughout the duration of the study
* Willing and able to make diet/lifestyle modifications in response to CGM data
* Able to read and understand English
* Able to attend study visits and complete the requirements of study

Exclusion Criteria:

* Currently taking or planning to take any form of insulin, sulfonylureas, meglitinides, or other anti-hyperglycemic diabetes medication that carry a known hypoglycemia risk
* Has used a personal CGM in the 90 days prior to consent
* Known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin
* Skin conditions that are not compatible with CGM wear
* Intended use of > 4g acetaminophen/day or hydroxyurea during the study
* Planning to become pregnant; pregnant; or lactating
* Current participation in another interventional clinical trial
* Unsuitable for participation due to any other cause, including but not limited to significant comorbidities, as determined by Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Phase 1 CGM-derived time in range (TIR) | From baseline (day -11 to day 0) to post-intervention (day 40 to day 50)
  % time with glucose 70-180 mg/dL is a core CGM metric; it will be assessed between groups and will be described as the 24-hour period, daytime period (6AM to 11:59PM), and nighttime period (12AM to 5:59PM)

SECONDARY OUTCOMES:
Total healthy eating index (HEI) score | Post-intervention period (day 40 to day 50)
  The total Healthy Eating Index is a measure of diet quality, independent of quantity, used to assess alignment of food intake with the Dietary Guidelines for Americans. HEI will be calculated using standard methods. A total score of 100 is possible. Higher scores indicate higher quality diets (better nutritional intake). Differences between groups during the post-intervention period will be described.

OTHER OUTCOMES:
CGM derived % time above >180 mg/dL | From baseline (day -11 to day 0) to post-intervention (day 40 to day 50)
  % time above >180 mg/dL is considered a core CGM metric; time above range. This will be described as the 24-hour period, daytime period (6AM to 11:59PM), and nighttime period (12AM to 5:59PM)
CGM-derived % time above >250 mg/dL | From baseline (day -11 to day 0) to post-intervention (day 40 to day 50)
  % time above >250 mg/dL is considered a core CGM metric; time above range. This will be described as the 24-hour period, daytime period (6AM to 11:59PM), and nighttime period (12AM to 5:59PM).
CGM-derived % time below <70 mg/dL | From baseline (day -11 to day 0) to post-intervention (day 40 to day 50)
  CGM-derived % time <70 mg/dL is considered a core CGM metric; time below range This will be described as the 24-hour period, daytime period (6AM to 11:59PM), and nighttime period (12AM to 5:59PM)
CGM-derived % time in tight range (% time with glucose 70-140 mg/dL) | From baseline (day -11 to day 0) to post-intervention (day 40 to day 50)
  Time in tight range is considered another CGM metric. This will be described as the 24-hour period, daytime period (6AM to 11:59PM), and nighttime period (12AM to 5:59PM).
% of participants reaching CGM-derived consensus targets | From baseline (day -11 to day 0) to post-intervention (day 40 to day 50)
  Consensus targets include the % of participants who reach >70% TIR (% time with glucose 70-180 mg/dL) and the % who reach ≥5% improvement in TIR (% time with glucose 70-180 mg/dL)
Total energy intake | From baseline (day -11) to post-intervention (day 40 to day 50)
  Energy intake will be calculated using 24 hour dietary recalls
Macronutrient intake | From baseline (day -11) to post-intervention (day 40 to day 50)
  Macronutrient intake will be calculated using 24 hour dietary recalls
Micronutrient intake | From baseline (day -11) to post-intervention (day 40 to day 50)
  Select micronutrient intake will be calculated using 24 hour dietary recalls
Diabetes Distress Scale-17 score | From baseline (day -11) to post-intervention (day 50)
  Diabetes distress will be measured using validated survey
HbA1c | From baseline (day -11) to post-intervention (day 50)
  HbA1c will be evaluated using point of care assessment
Body weight | From baseline (day -11) to post-intervention (day 50)
  Body weight based on calibrated study scale
Body mass index (BMI) | From baseline (day -11) to post-intervention (day 50)
  kg/m2 will be used to calculate BMI
Fidelity to the intended intervention | Post-intervention period (day 40 to day 50)
  Survey of care providers and participants will assess: dose (minutes of intervention), content (were intended intervention components delivered), perception of content enactment and satisfaction with intervention
Patient-reported behavioral change | Post-intervention period (day 40 to day 50)
  Survey of patient's perception of behavior change during the intervention to help describe mechanisms that may explain study results
Phase 2 CGM-derived time in range (TIR) | From post-intervention (day 40 to day 50) to follow-up (day 170 to day 180)
  % time with glucose 70-180 mg/dL from post-intervention to 4-month follow-up for combined NFA and SDA arms.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Willis, PhD, Principal Investigator — HealthPartners Institute, International Diabetes Center
Locations (1):
- HealthPartners Institute dba International Diabetes Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
As allowable by the governing IRB and organizational legal requirements, select, de-identified datasets for the completed project will be made available. All datasets will be shared in compliance with human subject protection and Health Insurance Portability and Accountability Act (HIPAA) privacy regulations. Platform for sharing will be determined at study close.